CLINICAL TRIAL: NCT02324530
Title: Evaluation of CPAP (Continuous Positive Airway Pressure) in the Planning of Radiation Treatments for Lung, Upper Abdomen and Left Breast Cancers
Brief Title: Evaluation of Continuous Positive Airway Pressure for Tumor Motion Management in Radiotherapy
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Principal Investigator, Dr. Zvi Symon MD, Chairman Radiation Oncology, Sheba Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMC-13-0637
Record Dates: First submitted 2014-12-10; First posted 2014-12-24 (Estimated); Last update posted 2014-12-24 (Estimated); Status verified 2014-12

CONDITIONS: Tumor Motion; "Continuous Positive Airway Pressure"; Lung Cancer; Breast Cancer; Abdominal Tumors
MeSH Terms: conditions — Lung Neoplasms; Breast Neoplasms; Abdominal Neoplasms | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Lung tumors (Experimental): Patients with > 1 cm tumor motion simulated using 4DCT with and without CPAP
  Interventions: Device: Continuous positive airway pressure (CPAP)
- Left sided Breast cancer (Experimental): Patients with heart abutting chest wall will be simulated using 4DCT with and without CPAP
  Interventions: Device: Continuous positive airway pressure (CPAP)
- Abdominal tumors (Experimental): Patient with liver metastases for SBRT or pancreatic tumors will be simulated using 4DCT with and without CPAP
  Interventions: Device: Continuous positive airway pressure (CPAP)

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP) — CT simulation with and without CPAP

SUMMARY:
This is a clinical study on patients to compare the effects of CPAP on lung volume diaphragm motion, heart position and tumor motion compared to free breathing. Only patients with significant tumor motion of greater than 1 cm amplitude or unfavorable chest wall geometry (heart close to chest wall) identified on standard imaging and simulation will be candidates for the study. Patients will be re- simulated and planned for radiation treatments with CPAP. The radiation plans generated with and without CPAP will be compared to evaluate the impact of CPAP on tumor motion and dose delivered to adjacent critical structures such as the heart and lung.

DETAILED DESCRIPTION:
Primary Objectives

* Evaluate effectiveness of CPAP to reproducibly reduce tumor and organ motion during radiation therapy treatments.
* Determine if CPAP allows for a reduction in normal tissue receiving radiation in chest and abdomen tumors and reduce heart exposure for patients receiving left breast irradiation.

Entry Criteria: This is a proof of concept and feasibility study. We propose to study 10 patients in each group for a total of thirty patients.

Eligibility criteria Group1. Lung tumors and nodules with tumor motion greater than 1 cm on standard imaging (n=10) Group2. Left sided breast tumors with unfavorable anatomy, viz heart abutting chest wall (n=10) Group3. Upper abdominal tumors: Liver and Pancreas with tumor motion greater than 1 cm. (n=10)

Pretreatment evaluations/management for patients meeting eligibility criteria CPAP All patients will be evaluated by a pulmonologist for their respiratory performances including physical examination, oxygen saturation and pulmonary function tests including DLCO that will serve for baseline measures. Then, adjustment session will be performed aiming to get adjusted to a CPAP device till the maximal tolerated pressure is not more than 16 cmH20 (TBD) for 30 minutes.

All patients must be able to tolerate CPAP and comply with daily treatment. 4D CT: CT simulation is the basis of conformal treatment planning [24, 25]. By using a slow acquisition time of 3 minutes the motion effects due to breathing can be captured and a 4D image generated. The tumor position can be imaged throughout the breathing cycle and a Maximum Intensity Projection (MIP) can be constructed and used in treatment planning. If there is no tumor motion the size of the MIP would equal the tumor size. The MIP size will increase with increasing tumor motion. The planning software allows us to calculate the MIP dimensions and volume. In addition total lung volumes and change in diaphragm position can be calculated (Figure 1). Radiation therapy planning parameters and volumetric analysis of tumor and normal tissue motion and position are calculated using available software and transferred to the Eclipse treatment planning system [17].

Treatment Planning:

The Eclipse treatment planning system will be used to generate and compare plans for treatment with and without CPAP.

Details of Intervention

Simulation All treatment planning and CPAP evaluation will be done in the radiation therapy department. Patients will be simulated on the Phillips 4D big bore CT simulator. The 4D scan which is done slowly over several minutes allows us to assess the full range of tumor motion throughout the respiratory cycle. An ITV is calculated which includes the actual tumor size with an expansion to account for the range of motion of the tumor by accounting for tumor location throughout the respiratory cycle (MIP) The MIP is the basis for the ITV and is the structure used for treatment planning. Patients recruited for the study will be re-simulated with the patient in the same position while undergoing CPAP treatment. ITV size and volume will be calculated for the tumor in in both the standard and CPAP studies and used for planning.

RPM: Diaphragm motion and respiratory cycle information will be obtained using the RPM for both the standard and the CPAP simulations. Differences in the respiratory wave cycle will be recorded [17].

The MIP/ITV images will be transferred to the Eclipse treatment planning system and using both the standard breathing and CPAP simulations treatment plans will be generated. Standard radiation plan evaluation parameters will be used and plans compared with respect to tumor coverage and normal tissue and normal tissue in the radiation field.

Radiation Plan:

Identical field arrangements will be generated for CPAP and non CPAP plans. Plans will be evaluated using standard radiation therapy planning parameters including: MIP or ITV, total lung volume, volume of GTV/CTV/PTV/ V20 and MLD.

Pre treatment Compare standard conformal radiation plans using Eclipse treatment planning system for each patient with and without CPAP.

RPM tracings with and without CPAP will be compared for all groups pre- treatment.

ELIGIBILITY:
Inclusion Criteria:

* Lung tumors and nodules with tumor motion greater than 1 cm on standard imaging
* Left sided breast tumors with unfavorable anatomy, viz heart abutting chest wall
* Upper abdominal tumors: Liver and Pancreas with tumor motion greater than 1 cm. (n=10)

Exclusion Criteria:

* Under 18 years old
* Inability to sign informed consent
* Pregnancy,
* Mental Illness,
* Not legally competent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-12; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in amplitude of tumor motion | 2 months
  Measurement of the Internal Target Volume in cc

SECONDARY OUTCOMES:
Reduction of radiation dose to critical organs | 2 months
  Mean Lung dose, Mean Heart dose measured in Gy

OTHER OUTCOMES:
Tolerability of CPAP | immediate
  Percentage of patients who tolerate CPAP

CONTACTS AND LOCATIONS:
Overall Officials: Zvi Symon, MD, Principal Investigator — Sheba Medical Center; Jeffrey Goldstein, MD, Principal Investigator — Sheba Medical Center; Yaacov R Lawrence, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba_Medical_Center, Tel Litwinsky, Israel